CLINICAL TRIAL: NCT02347423
Title: Immunogenicity and Safety of 3 Adjuvated Reduced Dose Inactivated Polio Vaccines (IPV-Al SSI) and Non-adjuvated Full Dose IPV SSI, Given as Primary Vaccinations to Infants at 6, 10 and 14 Weeks of Age
Brief Title: 3 Adjuvated Reduced Dose IPV-Al SSI and Non-adjuvated Full Dose IPV SSI Given as Primary Vaccinations to Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Quintiles, Inc. (Industry); Larix A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VIPV-05; 2014-003449-88 (EudraCT Number)
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Poliomyelitis
Keywords: Poliomyelitis immunization; primary series
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1/3 IPV-Al SSI (Experimental): 3 vaccinations of 1/3 IPV-Al SSI given at 6, 10 and 14 weeks of age
  Interventions: Biological: Primary series of immunisation comprised by 3 vaccinations IPV-Al SSI
- 1/5 IPV-Al SSI (Experimental): 3 vaccinations of 1/5 IPV-Al SSI given at 6, 10 and 14 weeks of age
  Interventions: Biological: Primary series of immunisation comprised by 3 vaccinations IPV-Al SSI
- 1/10 IPV-Al SSI (Experimental): 3 vaccinations of 1/10 IPV-Al SSI given at 6, 10 and 14 weeks of age
  Interventions: Biological: Primary series of immunisation comprised by 3 vaccinations IPV-Al SSI
- IPV Vaccine SSI (Active Comparator): 3 vaccinations of IPV Vaccine SSI given at 6, 10 and 14 weeks of age, The comparator IPV Vaccine SSI contains: Type 1: 40DU, Type 2: 8 DU and Type 3: 32 DU.
  Interventions: Biological: IPV Vaccine SSI

INTERVENTIONS:
Biological: Primary series of immunisation comprised by 3 vaccinations IPV-Al SSI
  Arms: 1/10 IPV-Al SSI; 1/3 IPV-Al SSI; 1/5 IPV-Al SSI
Biological: IPV Vaccine SSI
  Arms: IPV Vaccine SSI

SUMMARY:
The background of the present clinical trial is the overall aim of the World Health Organization (WHO) to obtain eradication of polio in the world. As part of this overall plan, inactivated polio vaccine (IPV) against poliovirus types 1, 2 and 3, at an affordable price, needs to be available in low resource third world countries. The intention of the present phase II clinical trial is to determine if reduced dose(s) of IPV-Al SSI are safe in the target population and do not decrease the immunogenicity clinically significantly compared to full dose IPV Vaccine SSI. The infants will receive three doses of one of the trial vaccines according to the WHO Expanded Program on Immunization (EPI) schedule of 6, 10 and 14 weeks of age.

A total of 824 healthy infants will be included in the trial.

DETAILED DESCRIPTION:
The trial is a phase II, dose investigation, parallel and multi-group, observer-blind, randomised, controlled, multicentre and non-inferiority trial.

Three investigational reduced dose adjuvated IPV-Al SSI vaccines and full dose IPV SSI vaccine will be investigated in four parallel groups:

* 1/3 IPV-Al SSI
* 1/5 IPV-Al SSI
* 1/10 IPV-Al SSI
* IPV Vaccine SSI (comparator)

At Visit 1 (screening and 1st vaccination visit), written informed consent is obtained and the subject's eligibility is assessed according to the pre-specified in-/exclusion criteria, including measurement of axillary temperature. If the subject is included, a pre-vaccination blood sample is taken for polio antibody determinations, and the subject is randomly allocated into one of the four groups to be vaccinated.

The subject is observed for ½ an hour after the injection of the investigational medical product (IMP) and any immediate adverse events observed are to be recorded. A diary, thermometer and ruler are handed out to the parents/guardians so that they can measure daily the injection site reactions and the axillary temperature the first 3 days and record any adverse event until the next visit.

At Visit 2 (2nd vaccination visit), 28-42 days after Visit 1, contraindications are reviewed, the 2nd vaccination is given, the diary is collected and adverse events and concomitant medications are recorded in the eCRF. A new diary is handed out.

At Visit 3 (3rd vaccination and blood sample visit), 28-42 days after Visit 2, a blood sample for immunogenicity assessment is taken, contraindications are reviewed, the 3rd vaccination is given, the diary is collected and adverse events and concomitant medications are recorded in the eCRF. A new diary is handed out.

At Visit 4 (blood sample visit), 28-42 days after Visit 3, a blood sample for immunogenicity assessment is taken, the diary is collected, and adverse events and concomitant medications are recorded in the eCRF. The trial termination form is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Infants of 6 weeks of age (+7 days) on date of first vaccination
2. Healthy assessed from medical history and physical examination
3. One parent/guardian has been properly informed about the trial and has signed the informed consent form
4. One parent/guardian grants access to the infant's trial related medical records
5. One parent/guardian is likely to comply with trial procedures

Exclusion Criteria:

1. Vaccinated with poliovirus vaccine (OPV or IPV), other than the trial vaccines, prior to inclusion or planned during the trial (e.g. on national polio immunisation days)
2. OPV vaccination or known exposure to poliovirus in household (living together) within 3 month prior to inclusion or planned during the trial
3. Has a sibling who is ≤5 years of age, and for whom OPV vaccination is planned during the trial
4. Low birth weight (< 2,500 g)
5. Known or suspected immunodeficiency (e.g. HIV, leukaemia, lymphoma) or family history of congenital or hereditary immunodeficiency
6. Severe uncontrolled chronic disease (e.g. neurologic, pulmonary, gastrointestinal, hepatic, renal or endocrine)
7. Known or suspected allergy to vaccine constituents (e.g. hypersensitivity to formaldehyde)
8. Acute severe febrile illness at day of vaccination deemed by the investigator to be a contraindication for vaccination
9. Uncontrolled coagulopathy or blood disorder contraindicating intramuscular injections or blood sampling
10. Treatment with a product which is likely to modify the immune response (e.g. blood products and immunoglobulins) prior to inclusion or planned during the trial
11. Participating in another clinical trial
12. Not suitable for inclusion in the opinion of the investigator

Ages: 42 Days to 49 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 824 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09-26 (Actual)

PRIMARY OUTCOMES:
For each of the 3 poliovirus types 1, 2 and 3, for the IPV-Al and IPV Vaccine SSI vaccines to evaluate: Type specific seroconversion rates based on baseline and 4 weeks post 3rd vaccincation | Change from baseline to 4 weeks post 3rd vaccincation

SECONDARY OUTCOMES:
Type-specific geometric mean titers (GMTs) | 4 weeks post 3rd vaccination for each vaccine
Type-specific seroprotection rates (titers ≥ 1/8) | 4 weeks post 3rd vaccination for each vaccine
Type-specific reverse cumulative titer distribution curves based on pre-vaccination and 4 weeks post 3rd vaccination serum titers for each vaccine | 4 weeks post 3rd vaccination for each vaccine
Adverse events following the vaccinations for each vaccine | From inclusion to 4 weeks post 3rd vaccincation

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Kromann, Study Director — Statens Serum Institut
Locations (1):
- Hospital Maternidad Nuestra de la Altagracia, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rivera L, Pedersen RS, Pena L, Olsen KJ, Andreasen LV, Kromann I, Nielsen PI, Sorensen C, Dietrich J, Bandyopadhyay AS, Thierry-Carstensen B. Immunogenicity and safety of three aluminium hydroxide adjuvanted vaccines with reduced doses of inactivated polio vaccine (IPV-Al) compared with standard IPV in young infants in the Dominican Republic: a phase 2, non-inferiority, observer-blinded, randomised, and controlled dose investigation trial. Lancet Infect Dis. 2017 Jul;17(7):745-753. doi: 10.1016/S1473-3099(17)30177-9. Epub 2017 Apr 25. PMID 28454674